CLINICAL TRIAL: NCT07180784
Title: Mindfulness-Based Stress Reduction Compared With Cognitive Behavioral Therapy to Improve Sleep and Mental Health in University Students With Insomnia
Brief Title: Psychological Interventions for Students With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Amélie Vézina, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-228 A-1 R-1
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: Insomnia; Mindfulness; Cognitive-behavior therapy; Students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled noninferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness based stress reduction (MBSR) (Experimental): The participants randomized to this arm received the 8-week MBSR program.
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)
- Cognitive Behaviour Therapy for Insomnia (CBT-I) (Active Comparator): The participants randomized to this arm received the 8-week CBT-I treatment.
  Interventions: Behavioral: Cognitive Behaviour Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — An intervention group offered to students that teaches meditation and yoga techniques, stress physiology, and mindfulness practices. Each group includes 5-6 participants and met once a week for 1.5 hours over a period of 8 consecutive weeks.
  Arms: Mindfulness based stress reduction (MBSR)
Behavioral: Cognitive Behaviour Therapy for Insomnia (CBT-I) — Traditional CBT-I was offered in small group sessions of 5 to 6 participants and lasted 1.5 hours each. They were held once a week over a period of 8 consecutive weeks.
  Arms: Cognitive Behaviour Therapy for Insomnia (CBT-I)

SUMMARY:
This study looked at university students who had trouble sleeping and compared two different programs designed to help with insomnia. One program was mindfulness-based stress reduction (MBSR), which focuses on meditation and awareness techniques, and the other was cognitive-behavioral therapy for insomnia (CBT-I), a structured approach that teaches strategies to change thoughts and habits around sleep. Participants were randomly assigned to one of the two programs. The researchers wanted to see how each program affected insomnia symptoms and related factors like stress, anxiety, mood, and overall quality of life. The researchers expected that CBT-I would lead to faster improvements right after the program, but they also believed that the mindfulness program would work just as well in the longer term, notably, three months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students aged 18 to 35 years from Université Laval;
* Meet the Diagnostic and Statistical Manual of Mental Disorders 5th Version (DSM-5) criteria for insomnia disorder;
* Report at least one consequence of insomnia on daytime functioning;
* Are available and committed to attending group therapy sessions of approximately 1.5 hours each, held over 8 consecutive weeks.

Exclusion Criteria:

* Presence of another major psychiatric disorder or other sleep disorder that could explain the insomnia symptoms;
* Presence of a serious medical condition (e.g., chronic pain);
* Previous participation in cognitive-behavioral therapy for insomnia (CBT-I) or prior completion of a mindfulness-based program (e.g., mindfulness-based stress reduction [MBSR], mindfulness-based cognitive therapy [MBCT]);
* Refusal to discontinue the use of substances (e.g., over-the-counter sleep aids, marijuana, alcohol) for the sole purpose of sleep aids for the duration of the study;
* Having a highly irregular sleep schedule (e.g., going to bed almost every night after 1:00 a.m. and waking up after 10:00 a.m.).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline: One week prior to the start of the 8-week program; Post-treatment: Within one day after completion of the 8-week program; Follow-up: Three months after completion of the 8-week program
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire used to evaluate the severity of insomnia symptoms (e.g., difficulties falling asleep). Total scores range from 0 to 28, with higher scores indicating greater insomnia severity (worse outcome). Score interpretation: 0-7 = no clinically significant insomnia; 8-14 = subthreshold insomnia; 15-21 = clinical insomnia (moderate severity); 22-28 = clinical insomnia (severe).

SECONDARY OUTCOMES:
The Patient Health Questionnaire-9 (PHQ-9) | Baseline: One week prior to the start of the 8-week program; Post-treatment: Within one day after completion of the 8-week program; Follow-up: Three months after completion of the 8-week program
  The Patient Health Questionnaire-9 (PHQ-9) is a nine-item self-report questionnaire used to assess the severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms (i.e., a worse outcome).
The Generalized Anxiety Disorder-7 (GAD-7) | Baseline: One week prior to the start of the 8-week program; Post-treatment: Within one day after completion of the 8-week program; Follow-up: Three months after completion of the 8-week program
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire used to assess the severity of generalized anxiety symptoms. Total scores range from 0 to 21, with higher scores indicating greater anxiety severity (worse outcome). Score interpretation: 0-4 = minimal anxiety; 5-9 = mild anxiety; 10-14 = moderate anxiety; 15-21 = severe anxiety.
The Perceived Stress Scale (PSS-14) | Baseline: One week prior to the start of the 8-week program; Post-treatment: Within one day after completion of the 8-week program; Follow-up: Three months after completion of the 8-week program
  The Perceived Stress Scale (PSS-14) is a 14-item self-report questionnaire that measures the degree to which individuals perceive their life situations as stressful over the past month. Total scores range from 0 to 56, with higher scores indicating greater perceived stress (worse outcome). Score interpretation: 0-13 = low stress; 14-26 = moderate stress; 27-40 = high stress.
The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Baseline: One week prior to the start of the 8-week program; Post-treatment: Within one day after completion of the 8-week program; Follow-up: Three months after completion of the 8-week program
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16-item self-report questionnaire that assesses overall satisfaction and enjoyment across various areas of daily functioning and quality of life. Total raw scores range from 14 to 70, which are typically converted into a percentage of the maximum possible score. Higher scores indicate greater enjoyment and satisfaction with quality of life (better outcome).

OTHER OUTCOMES:
Actigraphy | Baseline: 10 days recording prior to the start of the 8-week program; Post-treatment: 10 days recording starting within one day after completion of the 8-week program
  The actigraph (Actiwatch 2, Philips Respironics, Bend, OR) is a wrist-worn device that measures movement to estimate sleep-wake patterns and activity levels over time. Data are typically reported as total sleep time, sleep onset latency, wake after sleep onset, and sleep efficiency. Higher sleep efficiency and longer total sleep time indicate better sleep outcomes, whereas longer sleep onset latency and greater wake after sleep onset indicate worse sleep outcomes.
Sleep diary | Baseline: 10 days recording prior to the start of the 8-week program; Post-treatment: 10 days recording within one day after completion of the 8-week program; Follow-up: 10 days recording three months after completion of the 8-week program
  The Sleep Diary is a daily self-report log used to record sleep patterns, bedtime habits, and related factors to better understand and manage sleep difficulties. Variables derived from the diary include total sleep time, sleep onset latency, wake after sleep onset, and sleep efficiency. Higher sleep efficiency and longer total sleep time indicate better sleep outcomes, whereas longer sleep onset latency and greater wake after sleep onset indicate worse sleep outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'étude des troubles du sommeil (CETS) de l'université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No